CLINICAL TRIAL: NCT05216432
Title: First-in-Human Study of Mutant-selective PI3Kα Inhibitor, RLY-2608, as a Single Agent in Patients With Advanced Solid Tumors and in Combination With Endocrine Therapy +/- a CDK4/6 or CDK4 Inhibitor in Patients With Advanced Solid Tumors or Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Relay Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RLY-2608-101
Record Dates: First submitted 2021-12-20; First posted 2022-01-31 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: PIK3CA Mutation; Solid Tumor, Adult; HER2-negative Breast Cancer; Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer; Unresectable Solid Tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; palbociclib; ribociclib

STUDY DESIGN:
Intervention Model Description: Single Agent Arm:
  Part 1(multiple ascending doses, QD or BID):unresectable or metastatic solid tumors with PIK3CA mutation per local assessment; Part 2 (RP2D determined in Part 1) Patients with unresectable or metastatic solid tumors with ≥1 PIK3CA mutation per local assessment will be enrolled protocol defined groups
  Double Combination Arm Part 1(multiple ascending doses, QD or BID): HR+, HER2- locally advanced or metastatic breast cancer with PIK3CA mutation per local assessment Part 2 (RP2D determined in Part 1) Group 1: patients who have not received prior PI3Kα inhibitor Group 2: patients who are intolerant to PI3Kα inhibitor
  Triple Combination Arms Part 1(multiple ascending doses, QD or BID): HR+, HER2- locally advanced or metastatic breast cancer with PIK3CA mutation per local assessment
  Part 2 (RP2D determined in Part 1) Patients with HR+, HER2-locally advanced or metastatic breast cancer with PIK3CA mutation per local assessment will be enrolled in protocol defined groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- RLY-2608 for patients with unresectable or metastatic solid tumors (Experimental): Multiple doses of RLY-2608 for oral administration.
  Interventions: Drug: RLY-2608
- RLY-2608 + fulvestrant combination for HR+ HER2- locally advanced or metastatic breast cancer (Experimental): Oral dose of RLY-2608 in addition to fulvestrant as determined during Part 1 Dose Escalation.
  Interventions: Drug: RLY-2608; Drug: Fulvestrant
- RLY-2608+fulvestrant+palbo125mg for HR+HER2- locally advanced metastatic breast cancer (Experimental): Oral dose of RLY-2608 in addition to fulvestrant and palbociclib 125mg as determined during Part 1 Dose Escalation.
  Interventions: Drug: RLY-2608; Drug: Fulvestrant; Drug: Palbociclib 125mg
- RLY-2608+fulvestrant+ribo400mg for HR+HER2- locally advanced metastatic breast cancer (Experimental): Oral dose of RLY-2608 in addition to fulvestrant and ribociclib 400mg as determined during Part 1 Dose Escalation.
  Interventions: Drug: RLY-2608; Drug: Fulvestrant; Drug: Ribociclib 400mg
- RLY-2608+fulvestrant+ribo600mg for HR+HER2- locally advanced metastatic breast cancer (Experimental): Oral dose of RLY-2608 in addition to fulvestrant and ribociclib 600mg as determined during Part 1 Dose Escalation.
  Interventions: Drug: RLY-2608; Drug: Fulvestrant; Drug: Ribociclib 600mg
- RLY-2608+fulvestrant+PF-07220060 100 mg for HR+ HER2- locally advanced or metastatic breast cancer (Experimental): Oral dose of RLY-2608 in addition to fulvestrant and PF-07220060 100 mg as determined during Part 1 Dose Escalation
  Interventions: Drug: RLY-2608; Drug: Fulvestrant; Drug: PF-07220060 100mg
- RLY-2608+fulvestrant+PF-07220060 300 mg for HR+ HER2- locally advanced or metastatic breast cancer (Experimental): Oral dose of RLY-2608 in addition to fulvestrant and PF-07220060 300 mg as determined during Part 1 Dose Escalation
  Interventions: Drug: RLY-2608; Drug: Fulvestrant; Drug: PF-07220060 300 mg

INTERVENTIONS:
Drug: RLY-2608 — RLY-2608 is a mutant-selective, oral PI3Kα inhibitor.
Drug: Fulvestrant — 500 mg fulvestrant is administered intramuscularly on Cycle 1 Day 1, Day 15, and Day 1 of each subsequent cycle (where a cycle is 28 days).
  Other Names: Faslodex
  Arms: RLY-2608 + fulvestrant combination for HR+ HER2- locally advanced or metastatic breast cancer; RLY-2608+fulvestrant+PF-07220060 100 mg for HR+ HER2- locally advanced or metastatic breast cancer; RLY-2608+fulvestrant+PF-07220060 300 mg for HR+ HER2- locally advanced or metastatic breast cancer; RLY-2608+fulvestrant+palbo125mg for HR+HER2- locally advanced metastatic breast cancer; RLY-2608+fulvestrant+ribo400mg for HR+HER2- locally advanced metastatic breast cancer; RLY-2608+fulvestrant+ribo600mg for HR+HER2- locally advanced metastatic breast cancer
Drug: Palbociclib 125mg — 125mg palbociclib is taken orally once daily for 28-day cycles that include 21 days of treatment followed by 7 days off treatment.
  Other Names: Ibrance
  Arms: RLY-2608+fulvestrant+palbo125mg for HR+HER2- locally advanced metastatic breast cancer
Drug: Ribociclib 400mg — 400mg ribociclib is taken orally once daily for 28-day cycles that include 21 days of treatment followed by 7 days off treatment.
  Other Names: Kisqali
  Arms: RLY-2608+fulvestrant+ribo400mg for HR+HER2- locally advanced metastatic breast cancer
Drug: Ribociclib 600mg — 600mg ribociclib is taken orally once daily for 28-day cycles that include 21 days of treatment followed by 7 days off treatment.
  Other Names: Kisqali
  Arms: RLY-2608+fulvestrant+ribo600mg for HR+HER2- locally advanced metastatic breast cancer
Drug: PF-07220060 100mg — PF-07220060 100 mg is taken orally twice daily at the same time with RLY-2608 during each 28-day cycle.
  Arms: RLY-2608+fulvestrant+PF-07220060 100 mg for HR+ HER2- locally advanced or metastatic breast cancer
Drug: PF-07220060 300 mg — PF-07220060 300 mg is taken orally twice daily at the same time with RLY-2608 during each 28-day cycle.
  Arms: RLY-2608+fulvestrant+PF-07220060 300 mg for HR+ HER2- locally advanced or metastatic breast cancer

SUMMARY:
This is an open-label, FIH study designed to evaluate the maximum tolerated dose, recommended Phase 2 dose, safety, tolerability, PK, pharmacodynamics, and preliminary antineoplastic activity of RLY-2608, in advanced solid tumor patients with a Phosphatidylinositol-4,5-bisphosphate-3 kinase, catalytic subunit alpha (PIK3CA) mutation in blood and/or tumor per local assessment. The study will evaluate RLY-2608 as a single agent for patients with unresectable or metastatic solid tumors. It will also evaluate RLY-2608 in combination RLY-2608 + fulvestrant and in triple combination RLY-2608 + fulvestrant + CDK4/6 inhibitor (palbociclib or ribociclib) or CDK4 inhibitor (PF-07220060) for patients with HR+ HER2- locally advanced or metastatic breast cancer. The RLY-2608 single agent arm, RLY-2608 + fulvestrant combination arm, and triple combination arms will have 2 parts: a dose escalation (Part 1) and a dose expansion (Part 2).

ELIGIBILITY:
Key Inclusion Criteria

Patient has ECOG performance status of 0-1

One or more documented primary oncogenic PIK3CA mutation(s) in blood and/or tumor per local assessment

Other potentially oncogenic PIK3CA mutations may be considered but must be approved by the Sponsor prior to enrollment.

Part 1 [Escalation] - Ability to provide archived tumor tissue or be willing to undergo pretreatment tumor biopsy to assess PIK3CA status retrospectively Part 2 [Expansion] - Submit tumor tissue prior to study drug initiation for determination of PIK3CA mutation retrospectively.

Key Inclusion for RLY-2608 Single Agent Arm

* [For Part 1: Escalation]: Evaluable disease per RECIST v1.1
* [For Part 2: Expansion]: Measurable disease per RECIST v1.1
* Disease that is refractory to standard therapy, intolerant to standard therapy, or has declined standard therapy.
* Part 1- histologically or cytologically confirmed diagnosis of unresectable or metastatic solid tumor
* Part 2 - Unresectable or metastatic solid tumor with PIK3CA mutation(s) and one of the following tumor types:

Group 1: clear cell ovarian cancer Group 2: head and neck squamous cell carcinoma Group 3: cervical cancer Group 4: other solid tumors, excluding colorectal, clear cell ovarian, head and neck squamous cell, and cervical cancers Group 5: unresectable or metastatic solid tumors with PIK3CA double mutations In addition, the SRC (with Sponsor approval) may choose to open additional group(s) of 20 participants to study the clinical activity, safety, and PK/PD with other specified solid tumor types.

Key Inclusion for Combination Arms:

* Doublet combination arms [Part 1 and Part 2]: Evaluable disease per RECIST v1.1
* Triplet combination arms:
* [Part 1 and Part 2 Dose Expansion, Group 1]: Evaluable disease per RECIST.
* [Part 2 Dose Expansion, Group 2]: Measurable disease per RECIST. Bone-only lytic or lytic/blastic disease with at least 1 measurable soft-tissue component per RECIST may be eligible.
* [For Part 1 and Part 2]: Male or female with histologically or cytologically confirmed diagnosis of HR+, HER2- unresectable or metastatic breast cancer that is not amenable to curative therapy. Females may be postmenopausal, premenopausal, or perimenopausal. Premenopausal or perimenopausal females must have a histologically or cytologically confirmed diagnosis of HR+ HER2- locally advanced or metastatic breast cancer that is not amenable to curative therapy and must have initiated treatment with a gonadotropin-releasing hormone (GnRH) agonist at least 4 weeks prior to start of study drug with continuation of GnRH agonist for the duration of study treatment (GnRH agonist recommended for males).
* Had previous treatment for breast cancer with: [Does not apply to triplet combination arms, Part 2 Dose Expansion, Group 2]:

  1. ≤1 line of chemotherapy in the metastatic setting
  2. ≥1 CDK4/6 inhibitor in either the adjuvant and/or metastatic setting
  3. ≥1 antiestrogen therapy in either adjuvant and/or metastatic setting, including, but not limited to, selective estrogen-receptor degraders (eg, fulvestrant), selective estrogen receptor modulators (eg, tamoxifen), and aromatase inhibitors (AI) (letrozole, anastrozole, exemestane), and
  4. ≥1 PARP inhibitor, if appropriate, if documented germline BRCA1/2 mutation Note: Systemic local, loco-regional, or adjuvant treatment with chemotherapy and PARP inhibitors is not to be included in enumeration or previous treatment

[For double combination arm; Part 2 Dose Expansion, Group 2]: Received prior treatment with a PI3Kα, AKT, or mTOR inhibitor and discontinued the inhibitor due to intolerance and not disease progression, where intolerance is defined as treatment discontinuation due to treatment related AE (eg. hyperglycemia, rash, diarrhea, stomatitis) other than severe hypersensitivity reaction and/or life-threatening reactions, such as anaphylaxis and Stevens-Johnson syndrome.

[For triple combination arms; Part 1 dose escalation]: Participants who had previous treatment for breast cancer with PI3Kα, AKT, mTOR inhibitors and discontiuned due to participant/physician decision, intolerance, or disease progression will be considered.

[For triple combination arms, Part 2 Dose Expansion, Group 2]: Participants must be intolerant to or have declined standard therapy for locally advanced or metastatic HR+/HER2- PIK3CA-mutated breast cancer. Prior endocrine therapy and CDK4/6inhibitors are allowed as follows:

1. Participants must have progressed during (neo)adjuvant endocrine therapy or within12 months of completing (neo)adjuvant endocrine therapy with an AI or tamoxifen.
2. If a CDK4/6 inhibitor was included as part of (neo)adjuvant therapy, disease must have recurred/progressed >12 months after completion of the CDK4/6 inhibitor portion of (neo)adjuvant therapy

Key Exclusion Criteria

Prior treatment with:

1. PI3Kα, AKT, or mTOR inhibitors (all arms except for doublet RLY-2608 + fulvestrant arm, Part 2, Group 2; and triplet combinations, Part 1 dose escalation).
2. Immune checkpoint inhibitors.
3. Triplet combinations RLY-2608 + CDK4 or CDK4/6 inhibitor + fulvestrant, Part 2 expansion, Group 2 only:

i. Prior systemic chemotherapy or antibody drug conjugate for locally advanced or metastatic disease. ii. Prior CDK2, CDK4, or CDK4/6 inhibitor as treatment for locally advanced or metastatic disease.

iii. Prior treatment with fulvestrant or any selective ER degrader, with the exception of patients who have received fulvestrant or any selective ER degrader as part of neoadjuvant therapy only and with treatment duration ≤6 months.

Type 1 or Type 2 diabetes requiring antihyperglycemic medication, or fasting plasma glucose ≥140 mg/dL and glycosylated hemoglobin (HbA1c) ≥7.0%.

History of allergy or hypersensitivity to any components or excipients of PI3K inhibitors. For combination arms only: allergy or hypersensitivity to any components or excipients of fulvestrant, palbociclib, ribociclib, and/or PF-07220060 as appropriate for the combination.

Past medical history of or ongoing ILD, or pneumonitis requiring intervention. Participants with past history of resolved Grade 1 pneumonitis may be considered, except in triple combination arms.

The following cardiac criteria:

* Mean resting corrected QT interval (QTc) >460 msec
* For triple combination arm with ribociclib: Mean QTcF ≥450 msec (this is what we confirmed is shown in the redacted version of the protocol.

CNS metastases or primary CNS tumor that is associated with progressive neurologic symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of RLY-2608 as a single agent | Cycle 1 (4-week cycle) of treatment for MTD and at the end of every cycle (4-week cycles) for RP2D until study discontinuation, approximately 24 months
Determination of maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of RLY-2608 in combination with fulvestrant | Cycle 1 (4-week cycle) of treatment for MTD and at the end of every cycle (4-week cycles) for RP2D until study discontinuation, approximately 24 months
Determination of maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of RLY-2608 in combination with fulvestrant and a CDK 4/6 inhibitor (palbociclib, ribociclib), and in combination with CDK4 inhibitor (PF-07220060) and fulvestrant | Cycle 1 (4-week cycle) of treatment for MTD and at the end of every cycle (4-week cycles) for RP2D until study discontinuation, approximately 24 months
Number of patients with adverse events and serious adverse events of RLY-2608 as a single agent | Every cycle (4-week cycles) until study discontinuation, approximately 24 months
Number of patients with adverse events and serious adverse events of RLY-2608 in combination with fulvestrant | Every cycle (4-week cycles) until study discontinuation, approximately 24 months
Number of patients with adverse events and serious adverse events of RLY-2608 in combination with fulvestrant and a CDK 4/6 inhibitor (palbociclib, ribociclib), and in combination with CDK4 inhibitor (PF-07220060) and fulvestrant | Every cycle (4-week cycles) until study discontinuation, approximately 24 months

SECONDARY OUTCOMES:
PIK3CA gene status in plasma circulating tumor deoxyribonucleic acid (ctDNA) and tumor tissue | Day 1 of Cycle 1 (each cycle is 28 days)
Pharmacokinetic parameters including maximum plasma drug concentration (Cmax) of RLY-2608 (and its metabolites, as appropriate) as single agent | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment, approximately 24 months
Pharmacokinetic parameters including area under the plasma concentration versus time curve during a dose interval (AUC0-tau) of RLY-2608 (and its metabolites, as appropriate) as single agent | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment, approximately 24 months
Pharmacokinetic parameters including half-life (t1/2) of RLY-2608 (and its metabolites, as appropriate) as single agent | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment, approximately 24 months
Pharmacokinetic parameters including maximum plasma drug concentration (Cmax) of RLY-2608 (and its metabolites, as appropriate) when RLY-2608 is administered in combination with fulvestrant | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment, approximately 24 months
Pharmacokinetic parameters including area under the plasma concentration versus time curve during a dose interval (AUC0-tau) of RLY-2608 (and its metabolites, as appropriate) when RLY-2608 is administered in combination with fulvestrant | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment, approximately 24 months
Pharmacokinetic parameters including half-life (t1/2) of RLY-2608 (and its metabolites, as appropriate) when RLY-2608 is administered in combination with fulvestrant | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment, approximately 24 months
PK parameters including maximum plasma drug concentration (Cmax) of RLY-2608 (and its metabolites, as appropriate) when RLY-2608 is administered in combination with fulvestrant + palbociclib or ribociclib, and in combination (PF-07220060) +fulvestrant | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment, approximately 24 months
PK parameters including area under the plasma concentration vs time curve during a dose interval (AUC0-tau) of RLY-2608 (and its metabolites, as appropriate) administered with fulvestrant + palbociclib, or ribociclib, or PF-07220060 | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment, approximately 24 months
Pharmacokinetic parameters including half-life (t1/2) of RLY-2608 (and its metabolites, as appropriate) when RLY-2608 is administered in combination with fulvestrant + palbociclib or ribociclib, and in combination with PF-07220060 +fulvestrant | Approximately every 2 weeks in Cycle 1 (4-week cycle) and every cycle through end of treatment, approximately 24 months
Changes in circulating blood of fasting glucose in RLY-2608 as a single agent | Approximately every week in Cycle 1 (4-week cycle), every two weeks in Cycle 2 (4-week cycle), and every cycle starting with Cycle 3 through end of treatment, approx 24 months
Changes in circulating blood of insulin in RLY-2608 as a single agent | Approximately every week in Cycle 1 (4-week cycle), every two weeks in Cycle 2 (4-week cycle), and every cycle starting with Cycle 3 through end of treatment, approx 24 months
Changes in circulating blood of C-peptide in RLY-2608 as a single agent | Approximately every week in Cycle 1 (4-week cycle), every two weeks in Cycle 2 (4-week cycle), and every cycle starting with Cycle 3 through end of treatment, approx 24 months
Changes in circulating blood of HbA1c in RLY-2608 as a single agent | Once in Cycle 2 (4-week cycle) and then once every 3rd cycle beginning with Cycle 5 through end of treatment, approximately 24 months
Changes in circulating blood of fasting glucose in RLY-2608 in combination with fulvestrant | Approximately every week in Cycle 1 (4-week cycle), every two weeks in Cycle 2 (4-week cycle), and every cycle starting with Cycle 3 through end of treatment, approx 24 months
Changes in circulating blood of insulin in RLY-2608 in combination with fulvestrant | Approximately every week in Cycle 1 (4-week cycle), every two weeks in Cycle 2 (4-week cycle), and every cycle starting with Cycle 3 through end of treatment, approx 24 months
Changes in circulating blood of C-peptide in RLY-2608 in combination with fulvestrant | Approximately every week in Cycle 1 (4-week cycle), every two weeks in Cycle 2 (4-week cycle), and every cycle starting with Cycle 3 through end of treatment, approx 24 months
Changes in circulating blood of HbA1c in RLY-2608 in combination with fulvestrant | Once in Cycle 2 (4-week cycle) and then once every 3rd cycle beginning with Cycle 5 through end of treatment, approximately 24 months
Changes in circulating blood of fasting glucose in RLY-2608 in combination with fulvestrant and a CDK4/6 inhibitor (palbociclib, ribociclib) and in combination with CDK4 inhibitor (PF-07220060) and fulvestrant | Approximately every week in Cycle 1 (4-week cycle), every two weeks in Cycle 2 (4-week cycle), and every cycle starting with Cycle 3 through end of treatment, approx 24 months
Changes in circulating blood of insulin in RLY-2608 in combination with fulvestrant and a CDK4/6 inhibitor (palbociclib, ribociclib), and in combination with CDK4 inhibitor (PF-07220060) and fulvestrant | Approximately every week in Cycle 1 (4-week cycle), every two weeks in Cycle 2 (4-week cycle), and every cycle starting with Cycle 3 through end of treatment, approx 24 months
Changes in circulating blood of C-peptide in RLY-2608 in combination with fulvestrant and a CDK4/6 inhibitor (palbociclib, ribociclib), and in combination with CDK4 inhibitor (PF-07220060) and fulvestrant | Approximately every week in Cycle 1 (4-week cycle), every two weeks in Cycle 2 (4-week cycle), and every cycle starting with Cycle 3 through end of treatment, approx 24 months
Changes in circulating blood of HbA1c in RLY-2608 in combination with fulvestrant and a CDK4/6 inhibitor (palbociclib, ribociclib), and in combination with CDK4 inhibitor (PF-07220060) and fulvestrant | Once in Cycle 2 (4-week cycle) and then once every 3rd cycle beginning with Cycle 5 through end of treatment, approximately 24 months
Objective response rate (ORR) as assessed by RECIST v1.1 | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Duration of Response (DOR) as assessed by RECIST v1.1 | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Disease Control Rate (DCR) as assessed by RECIST v1.1 | Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months
Clinical benefit rate (CBR) as assessed by RECIST v1.1 | [Time Frame: Approximately every 8 weeks during treatment and every 12 weeks after the last dose in the absence of progressive disease, approximately 36 months]

CONTACTS AND LOCATIONS:
Locations (37):
- United States (24):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of California-San Diego, San Diego, California
  - HealthONE, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Florida Cancer Specialists, Orlando, Florida
  - Boca Raton Clinical Research (BRCR) Global, Plantation, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Community Health Network, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine St. Louis, St Louis, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Rutgers University, New Brunswick, New Jersey
  - NYU Langone, New York, New York
  - Columbia University Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - University of Utah- Huntsman Cancer Center, Salt Lake City, Utah
  - Inova Schar Cancer Center, Fairfax, Virginia
  - NEXT Virginia, Fairfax, Virginia
  - UW Carbone Cancer Center, Madison, Wisconsin
- Australia (3):
  - St Vincents Hospital, Sydney, New South Wales
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- France (3):
  - Centre Léon Bérard, Lyon, Auvergne-Rhône-Alpes
  - Institute Bergonié, Bordeaux
  - Gustave Roussy, Villejuif
- Istituto Europeo di Oncologia IRCCS, Milan, Italy
- Spain (6):
  - Vall d'Hebron Instituto de Oncologia, Barcelona, Barcelona
  - START Barcelona, Barcelona, Catalonia
  - Instituto Valenciano de Oncologia, Valencia, Valencia
  - Institut Catala D'Oncologia - Badalona (ICO Badalona), Barcelona
  - START Madrid - Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No